CLINICAL TRIAL: NCT05081479
Title: Phase I Study of N-Acetylcysteine to Optimize Metabolic Tumor Microenvironment in CD19 CAR T-cell Therapy in Lymphoma
Brief Title: A Study of N-Acetylcysteine (N-AC) in People Receiving CAR T-cell Therapy for Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-386
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma
Keywords: N-AC; N-Acetylcysteine; Lymphoma; CD19 CAR T-cell Therapy; 21-386; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants with Lymphoma, Cohort 1 (Experimental): The first dose escalation cohort in the study will be treated at 25% of that target dose level
  Interventions: Drug: N-Acetylcysteine
- Participants with Lymphoma, Cohort 2 (Experimental): The second cohort in the study will be treated at 50% of that target dose level
  Interventions: Drug: N-Acetylcysteine
- Participants with Lymphoma, Cohort 3 (Experimental): The third cohort in the study will be treated at 100% of that target dose level only if no DLTs are seen at lower doses.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — N-AC infusion will begin the day before CAR T cell infusion and continuously infused over 24-hours for 14 days or until time of discharge whichever is earlier. Interruptions of N-AC infusion for medical reasons are permissible. The dose for patients <45kg will be adjusted to weight based dosing.
  Other Names: N-AC

SUMMARY:
The purpose of this study is to test the safety of N-AC when given in combination with Yescarta to people with lymphoma. This study will test different doses of N-AC to find the highest dose that causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients who will receive axicabtagene ciloleucel for treatment of lymphoma
* Patients must have adequate end organ function to be eligible for this study as defined by the following criteria:

  * ECOG performance status 0-2
  * Hematologic function with ANC ≥ 1000, Hgb ≥ 8, Plt ≥ 50k unless there is disease related hematologic toxicity
  * Renal function with CrCr ≥ 40 ml/min or Cr ≤ 1.5 x ULN
  * Hepatic function with ALT/AST ≤ 2.5 x ULN, TBili ≤ 1.5 x ULN.

Exclusion Criteria:

* Patients with known allergy to N-AC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of N-AC | Up to 1 year
  This is a phase 1 dose escalation and expansion study to determine the maximum tolerated dose and recommended phase 2 dose of NAC given in conjunction with axicabtagene ciloleucel.

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org